CLINICAL TRIAL: NCT03167983
Title: The Gut-Brain Axis in Dementia: Biomarker and Novel Intervention Strategies
Brief Title: Microbiome and Dementia
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Demenz
Record Dates: First submitted 2017-05-15; First posted 2017-05-30 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dementia: patients with dementia
- control: healthy control

SUMMARY:
From this study, it is hoped to learn if and how the gut microbiome composition, gut permeability and inflammation in patients with dementia are associated with each other. Dysbiosis may lead to an increased gut permeability, bacterial translocation and inflammation which may influence pathogenesis and progression of dementia.

The novel aspect of the study will be to understand the association between gut microbiome composition, gut permeability and the presence of dementia. This will help to better understand the pathogenesis of dementia and lead to the development of novel therapeutic strategies. If this hypothesis holds true, the study will be the basis to develop new treatment options for dementia.

DETAILED DESCRIPTION:
Dementia is a disease that presents with deterioration in memory, thinking, behaviour and the ability to perform everyday activities. Worldwide 47.5 million people are affected and incidence of dementia is increasing. Dementia leads to disability and dependency among older people worldwide and thereby has a huge physical, psychological, social and economic impact on caregivers, families and society. Alzheimers disease (AD) is the most common form of dementia accounting for 60-70% of the cases; other forms include Lewy body dementia, frontotemporal dementia, vascular dementia and Parkinsons disease with dementia. In AD, pathologic protein aggregates of amyloid beta and hyperphosphorylated tangles of tau-protein which deposit as neurofibrillary tangles are typical features. This leads to neuroinflammation, mainly mediated by the innate immune system. The most important cells in this process are microglia cells, which represent the resident macrophages of the brain. Although microglia is able to remove extracellular amyloid beta, in later stages of the disease cells remain in a dystrophic state and cannot exert their beneficial functions. Microglia maturation and function is critically dependent on short-chain fatty acids produced by the gut microbiome and therefore highlights the microbiome as a potential diagnostic and therapeutic target in dementia.

The role of the commensal microbial population of the human body - especially the intestinal microbiome - in various diseases is emerging due to the development of advanced analysis techniques. Recently the concept of the gut brain-axis has been established. Several pathways including the autonomic nervous system, the enteric nervous system, the neuroendocrine system and the immune system allow a communication between gut and brain but may also be involved in disease development.

During ageing, the gut microbiome composition undergoes changes. A decrease in diversity, a loss of beneficial taxa and an increase of facultative pathogens has been described. Diet and the place of residence play an important role in the shaping of the microbiome. Aging is also associated with inflammation - often termed as "inflammaging" associated with an increase in gut permeability, mucosal inflammation and bacterial translocation.

Since the main risk factor for developing dementia, especially AD, is aging, it is very likely that the gut-brain axis is critically involved in dementia development.

Animal studies so far suggest that AD is associated with changes in the gut microbiome composition with a decrease in beneficial, anti-inflammatory genera. Furthermore, genetic alterations in amyloid genes can influence microbiome composition in mice, pointing towards a vicious cycle in AD development.

In humans, so far no studies on the gut microbiome composition in patients with dementia have been published. However, there is evidence that the composition of the microbiome in subgingival plaques is altered in dementia and associated with cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Age >18y
* Dementia (Alzheimer type and mixed type)
* Informed consent signed by the patient or his legal representative
* Mini Mental State Examination ≤ 26

Exclusion Criteria:

* Other forms of dementia
* Inflammatory bowel diseases
* Liver cirrhosis
* Antibiotic treatment within the last 14 days
* Any other condition or circumstance, which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol

Healthy controls

* Age >18y
* Informed consent
* No known acute or chronic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with dementia and age matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Alpha diversity | single measurement at baseline
  Chao1 index

SECONDARY OUTCOMES:
gut permeability | single measurement at baseline
  zonulin
bacterial translocation | single measurement at baseline
  serum biomarker of bacterial translocation
inflammation | single measurement at baseline
  serum biomarker of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stadlbauer V, Engertsberger L, Komarova I, Feldbacher N, Leber B, Pichler G, Fink N, Scarpatetti M, Schippinger W, Schmidt R, Horvath A. Dysbiosis, gut barrier dysfunction and inflammation in dementia: a pilot study. BMC Geriatr. 2020 Jul 20;20(1):248. doi: 10.1186/s12877-020-01644-2. PMID 32690030